CLINICAL TRIAL: NCT02514746
Title: Assessment of Long Term Immunogenicity of Japanese Encephalitis Live Attenuated SA-14-14-2 Vaccine in Previously Vaccinated Bangladeshi Children and Antibody Response and Safety to a Booster Dose
Brief Title: Long-term Immunogenicity After Receipt of JE Vaccine and Antibody Response and Safety to a Booster Dose
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: PATH (Other)
Collaborators: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: JEV07; PR-15036 (Other: International Centre for Diarrhoeal Disease Research, Bangladesh)
Record Dates: First submitted 2015-07-15; First posted 2015-08-04 (Estimated); Results first posted 2020-10-19 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-08

CONDITIONS: Encephalitis, Japanese
Keywords: Japanese Encephalitis Vaccines; Flavivirus Infections
MeSH Terms: conditions — Encephalitis, Japanese; Flavivirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Live Attenuated JE SA-14-14-2 Vaccine (CD-JEV) (Experimental): Participants previously vaccinated with CD-JEV will receive a booster dose of live, attenuated Japanese encephalitis SA-14-14-2 vaccine four years after initial vaccination.
  Interventions: Biological: Live Attenuated Japanese Encephalitis SA-14-14-2 Vaccine

INTERVENTIONS:
Biological: Live Attenuated Japanese Encephalitis SA-14-14-2 Vaccine — 0.5 mL subcutaneous injection
  Other Names: CD-JEV; CD.JEVAX®; RS.JEV®

SUMMARY:
This study aims to understand the persistence of the Japanese encephalitis (JE) antibody response in previously vaccinated children. The proposed study will enrol Bangladeshi children who had previously participated in a lot to lot consistency study (JEV05; NCT01567865) of JE live attenuated SA 14-14-2 vaccine (CD-JEV).

DETAILED DESCRIPTION:
Study participants previously immunized with CD-JEV (Clinical Trials identifier: NCT01567865, JEV05) will have serum collected three and four years after initial vaccination to assess long-term immunogenicity. Four years after receiving the initial dose of CD-JEV, eligible participants will be vaccinated with a second subcutaneous dose of CD-JEV to assess the antibody response.

Participants will be monitored for safety for 28 days following receipt of the booster dose.

ELIGIBILITY:
Inclusion Criteria:

* Participant in JEV05 study (NCT01567865) and received one dose of CD-JEV.
* Resides in the Matlab or Mirpur study area.
* At least one parent or guardian willing to provide written informed consent.

Exclusion Criteria:

* Received a second dose of Japanese encephalitis vaccine within the past three years.
* Received immunoglobulins and/or any blood products within 90 days prior to enrollment.
* Been diagnosed with a primary or acquired immunodeficiency, including human immunodeficiency virus (HIV) infection within the past three years.

Ages: 43 Months to 51 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 561 (Actual)
Dates: Start 2015-07-30 (Actual); Primary Completion 2016-12-15 (Actual); Study Completion 2017-01-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: K Zaman, PhD, MPH, MBBS, Principal Investigator — International Centre for Diarrhoeal Disease Research, Bangladesh

REFERENCES:
- [Result] Zaman K, Naser AM, Power M, Yaich M, Zhang L, Ginsburg AS, Luby SP, Rahman M, Hills S, Bhardwaj M, Flores J. Lot-to-lot consistency of live attenuated SA 14-14-2 Japanese encephalitis vaccine manufactured in a good manufacturing practice facility and non-inferiority with respect to an earlier product. Vaccine. 2014 Oct 21;32(46):6061-6. doi: 10.1016/j.vaccine.2014.09.012. Epub 2014 Sep 18. PMID 25239483
- [Derived] Zaman K, Yunus M, Aziz AB, Feser J, Mooney J, Tang Y, Ellison DW, Thaisomboonsuk B, Zhang L, Neuzil KM, Marfin AA, Letson GW. Antibody persistence and immune memory response following primary vaccination and boosting with live attenuated SA 14-14-2 Japanese encephalitis vaccine (CD-JEV) in Bangladesh: A phase 4 open-label clinical trial. Vaccine X. 2022 Feb 5;10:100143. doi: 10.1016/j.jvacx.2022.100143. eCollection 2022 Apr. PMID 35243320

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study enrolled Bangladeshi children who had participated in Study JEV05 (NCT01567865) and received a single dose of live attenuated Japanese encephalitis vaccine (CD-JEV).
  The first visit in this study was 3 years after vaccination in JEV05. At the 2nd study visit, 4 years after initial vaccination, children received a booster dose of CD-JEV.
Pre-assignment Details: Children were analyzed based on whether they received vaccine from the new or old facility in Study JEV05:
  * Group A: Received CD-JEV from new facility in Study JEV05
  * Group B: Received CD-JEV from old facility in Study JEV05
Groups:
- Group A: CD-JEV: Participants previously vaccinated with CD-JEV manufactured in the new facility received a booster dose of live, attenuated Japanese encephalitis SA-14-14-2 vaccine by subcutaneous injection four years after initial vaccination.
- Group B: CD-JEV: Participants previously vaccinated with CD-JEV manufactured in the old facility received a booster dose of live, attenuated Japanese encephalitis SA-14-14-2 vaccine by subcutaneous injection four years after initial vaccination.
Period: Overall Study
Arm/Group | Group A: CD-JEV | Group B: CD-JEV
Started (All enrolled participants) | 437 | 124
Valid Serology 3 Years Post Primary Dose | 437 | 123
Valid Serology 4 Years Post Primary Dose | 424 | 109
Received CD-JEV Booster Vaccine | 424 | 109
Completed (Completed all study visits through 28 days post booster vaccination.) | 415 | 109
Not Completed | 22 | 15
Not completed — Chronically Ill | 1 | 2
Not completed — Physician Decision | 4 | 2
Not completed — Withdrawal by Subject | 12 | 10
Not completed — Other | 5 | 1

BASELINE CHARACTERISTICS:
Population: All enrolled participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A: CD-JEV | Group B: CD-JEV | Total
Number analyzed (Participants) | 437 | 124 | 561
Age, Continuous [Mean (Standard Deviation); unit: months] | 47.7 (1.6) | 47.8 (1.4) | 47.7 (1.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 226 | 65 | 291
  Male | 211 | 59 | 270
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Bangladesh | 437 | 124 | 561

OUTCOME MEASURES:

1. Primary Outcome: Seroprotection Rate Three and Four Years After Initial Vaccination With CD-JEV
Description: Seroprotection rate is defined as the percentage of participants with an anti-Japanese encephalitis (JE) neutralizing antibody titer ≥ 1:10 as measured using a 50% plaque reduction neutralization test (PRNT-50). Seroprotection was assessed at 3 and 4 years after the initial vaccination in Study JEV05, prior to participants receiving a booster vaccination in the current study.
Time Frame: 3 years after initial vaccination (Study Day 1) and 4 years after initial vaccination (Study Day 365)
Population: Enrolled participants with at least one serology result at Year 3 (Day 1) or Year 4 (Day 365), prior to receiving the booster dose (long-term assessment intention-to-treat population [ITT]).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Total: Participants previously vaccinated with CD-JEV received a booster dose of live, attenuated Japanese encephalitis SA-14-14-2 vaccine by subcutaneous injection four years after initial vaccination.
Arm/Group | Group A: CD-JEV | Group B: CD-JEV | Total
Number analyzed (Participants) | 437 | 123 | 560
percentage of participants
  Year 3 | 9.2 [6.8 to 12.2] | 9.8 [5.7 to 16.3] | 9.3 [7.2 to 12.0]
  Year 4: number analyzed (Participants) | 424 | 109 | 533
  Year 4 | 12.5 [9.7 to 16.0] | 11.9 [7.1 to 19.3] | 12.4 [9.9 to 15.5]
Statistical Analysis 1: Comparison: Group A: CD-JEV vs Group B: CD-JEV; Difference at Year 3; Test type: Other; Difference (Group A - B) = -0.6, 95% CI 2-sided [-7.5 to 4.5]
Statistical Analysis 2: Comparison: Group A: CD-JEV vs Group B: CD-JEV; Difference at Year 4; Test type: Other; Difference (Group A - B) = 0.6, 95% CI 2-sided [-7.4 to 6.5]

2. Primary Outcome: Geometric Mean Titer of Anti-JE Neutralizing Antibodies Three and Four Years After Initial Vaccination With CD-JEV
Description: The geometric mean titer (GMT) of anti-JE neutralizing antibodies 3 and 4 years after initial vaccination with CD-JEV in Study JEV05 and prior to receiving the booster vaccination in the current study, measured using PRNT-50.
Time Frame: 3 years after initial vaccination (Study Day 1) and 4 years after initial vaccination (Study Day 365)
Population: Enrolled participants with at least one serology result at Year 3 (Day 1) or Year 4 (Day 365), prior to receiving the booster dose.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Group A: CD-JEV | Group B: CD-JEV | Total
Number analyzed (Participants) | 437 | 123 | 560
titer
  Year 3 | 5.8 [5.5 to 6.1] | 5.8 [5.3 to 6.4] | 5.8 [5.6 to 6.1]
  Year 4: number analyzed (Participants) | 424 | 109 | 533
  Year 4 | 6.1 [5.8 to 6.5] | 6.0 [5.4 to 6.7] | 6.1 [5.8 to 6.4]
Statistical Analysis 1: Comparison: Group A: CD-JEV vs Group B: CD-JEV; Geometric mean titer ratio at Year 3; Test type: Other; GMT Ratio (Group A/B) = 1.0, 95% CI 2-sided [0.9 to 1.1]
Statistical Analysis 2: Comparison: Group A: CD-JEV vs Group B: CD-JEV; Geometric mean titer ratio at Year 4; Test type: Other; GMT Ratio (Group A/B) = 1.0, 95% CI 2-sided [0.9 to 1.1]

3. Secondary Outcome: Seroprotection Rate 7 Days and 28 Days After Booster Dose
Description: Seroprotection rate is defined as the percentage of study participants with an anti-JE neutralizing antibody titer ≥1:10 assessed using PRNT-50.
Time Frame: 7 days and 28 days following booster vaccination (Study Days 372 and 393)
Population: Participants who received the booster dose of CD-JEV and had at least one serology result 7 days or 28 days after the booster vaccination (ITT booster analysis set).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group A: CD-JEV | Group B: CD-JEV | Total
Number analyzed (Participants) | 417 | 109 | 526
percentage of participants
  7 days after booster: number analyzed (Participants) | 417 | 107 | 524
  7 days after booster | 90.6 [87.5 to 93.1] | 94.4 [88.3 to 97.4] | 91.4 [88.7 to 93.5]
  28 days after booster: number analyzed (Participants) | 415 | 109 | 524
  28 days after booster | 97.8 [95.9 to 98.9] | 99.1 [95.0 to 99.8] | 98.1 [96.5 to 99.0]
Statistical Analysis 1: Comparison: Group A: CD-JEV vs Group B: CD-JEV; Difference at 7 days post booster vaccination; Test type: Other; Difference (Group A - B) = -3.7, 95% CI 2-sided [-8.1 to 2.8]
Statistical Analysis 2: Comparison: Group A: CD-JEV vs Group B: CD-JEV; Difference at 28 days post booster vaccination; Test type: Other; Difference (Group A - B) = -1.3, 95% CI 2-sided [-3.3 to 3.0]

4. Secondary Outcome: GMT of Anti-JE Neutralizing Antibodies 7 Days and 28 Days After Booster Dose
Description: Geometric mean titer of anti-JE neutralizing antibodies measured using PRNT-50.
Time Frame: 7 days and 28 days following booster vaccination (Study Days 372 and 393)
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Group A: CD-JEV | Group B: CD-JEV | Total
Number analyzed (Participants) | 417 | 109 | 526
titer
  7 days after booster: number analyzed (Participants) | 417 | 107 | 524
  7 days after booster | 98.8 [86.1 to 113.3] | 135.4 [105.7 to 173.5] | 105.4 [93.4 to 118.9]
  28 days after booster: number analyzed (Participants) | 415 | 109 | 524
  28 days after booster | 156.2 [140.6 to 173.4] | 215.4 [177.3 to 261.7] | 167.0 [152.2 to 183.2]
Statistical Analysis 1: Comparison: Group A: CD-JEV vs Group B: CD-JEV; Geometric mean titer ratio 7 days after booster dose; Test type: Other; GMT Ratio (Group A/B) = 0.7, 95% CI 2-sided [0.5 to 1.0]
Statistical Analysis 2: Comparison: Group A: CD-JEV vs Group B: CD-JEV; Geometric mean titer ratio 28 days after booster dose; Test type: Other; GMT Ratio (Group A/B) = 0.7, 95% CI 2-sided [0.6 to 0.9]

5. Secondary Outcome: Seroconversion Rate 7 Days and 28 Days After Booster Dose
Description: Seroconversion rate is defined as the percentage of study participants with either:
  * For participants who were seronegative at Baseline (defined as anti-JE neutralizing antibody titer of < 1:10 assessed using PRNT-50 at Year 4, prior to booster vaccination): A change in serostatus from seronegative (anti-JE neutralizing antibody titer of < 1:10) to positive (anti-JE neutralizing antibody titer ≥ 1:10)
  * For participants who were seropositive at Baseline (defined as an anti-JE neutralizing antibody titer ≥1:10 assessed using PRNT-50 at Year 4, prior to booster vaccination): a 4-fold increase in anti-JE neutralizing antibody titer relative to Baseline anti-JE neutralizing antibody titer
Time Frame: 7 days and 28 days following booster vaccination (Study Days 372 and 393)
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group A: CD-JEV | Group B: CD-JEV | Total
Number analyzed (Participants) | 417 | 109 | 526
percentage of participants
  7 days after booster: number analyzed (Participants) | 417 | 107 | 524
  7 days after booster | 88.7 [85.3 to 91.4] | 91.6 [84.8 to 95.5] | 89.3 [86.4 to 91.7]
  28 days after booster: number analyzed (Participants) | 415 | 109 | 524
  28 days after booster | 96.4 [94.1 to 97.8] | 98.2 [93.6 to 99.5] | 96.8 [94.9 to 98.0]
Statistical Analysis 1: Comparison: Group A: CD-JEV vs Group B: CD-JEV; Difference at 7 days post booster vaccination; Test type: Other; Difference (Group A - B) = -2.9, 95% CI 2-sided [-8.0 to 4.5]
Statistical Analysis 2: Comparison: Group A: CD-JEV vs Group B: CD-JEV; Difference at 28 days post booster vaccination; Test type: Other; Difference (Group A - B) = -1.8, 95% CI 2-sided [-4.4 to 3.0]

6. Secondary Outcome: GMT Ratio of Anti-JE Neutralizing Antibody Titers Between Post-Booster and Pre-Booster Vaccination
Description: To evaluate the magnitude of the increase in GMTs, the GMT ratio of anti-JE neutralizing antibody titers between post-booster vaccination and pre-booster vaccination was calculated for the following:
  * GMT of anti-JE neutralizing antibodies at 7 days after booster vaccination to the Year 4, pre-booster GMT of anti-JE neutralizing antibodies
  * GMT of anti-JE neutralizing antibodies at 28 days after booster vaccination to the Year 4, pre-booster GMT of anti-JE neutralizing antibodies
Time Frame: 4 years after the initial vaccination (Study Day 365, pre-booster vaccination) and 7 and 28 days following booster vaccination (Study Days 372 and 393)
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: ratio
Arm/Group | Group A: CD-JEV | Group B: CD-JEV | Total
Number analyzed (Participants) | 417 | 109 | 526
ratio
  7 days after booster: number analyzed (Participants) | 417 | 107 | 524
  7 days after booster | 16.2 [14.2 to 18.5] | 22.5 [17.5 to 28.9] | 17.3 [15.4 to 19.4]
  28 days after booster: number analyzed (Participants) | 415 | 109 | 524
  28 days after booster | 25.9 [23.3 to 28.7] | 35.9 [29.4 to 43.9] | 27.7 [25.3 to 30.4]

7. Secondary Outcome: Number of Participants With Immediate Reactions 30 Minutes Following Booster Vaccination
Description: The number of participants with at least one occurrence of an immediate reaction, including local, systemic, or unsolicited adverse event that occurred within 30 minutes of the booster vaccination.
Time Frame: 30 minutes following booster vaccination (Study Day 365)
Population: Participants who received the booster vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | Group A: CD-JEV | Group B: CD-JEV | Total
Number analyzed (Participants) | 424 | 109 | 533
Participants
  Any immediate reaction | 3 | 1 | 4
  Injection site pain | 1 | 0 | 1
  Injection site swelling | 3 | 1 | 4

8. Secondary Outcome: Number of Participants With Solicited Local Reactions Occurring Within 7 Days of Booster Vaccination
Description: Participants were monitored for local reactions from 30 minutes through 7 days post booster vaccination. Local reactions (at the injection site) included the following:
  * Ecchymosis (bruising)
  * Erythema (redness)
  * Edema (swelling)
  * Induration (hardness)
  * Pain/tenderness
  Local ecchymosis, erythema, edema, and induration were graded as follows:
  * Grade 1: ≤ 2.5 cm in diameter
  * Grade 2: > 2.5 cm in diameter with < 50% surface area of extremity involved
  * Grade 3: ≥ 50% surface area of extremity involved OR ulceration OR secondary infection OR phlebitis OR sterile abscess OR drainage
  * Grade 4: potentially life-threatening consequences
  Injection site pain/tenderness were graded as follows:
  * Grade 1: causing no or minimal limitation in use of limb
  * Grade 2: causing greater than minimal limitation of use of limb
  * Grade 3: causing inability to perform usual social or functional activities
  * Grade 4: inability to perform basic self-care OR hospitalization indicated.
Time Frame: From 30 minutes to 7 days following booster vaccination (Study Day 365 to 372)
Population: Participants who received the booster vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | Group A: CD-JEV | Group B: CD-JEV | Total
Number analyzed (Participants) | 424 | 109 | 533
Participants
  Any Local Reaction | 1 | 1 | 2
  Ecchymosis | 0 | 0 | 0
  Erythema | 0 | 0 | 0
  Edema | 0 | 0 | 0
  Induration | 0 | 0 | 0
  Pain/tenderness | 1 | 1 | 2
  Pain/tenderness - Grade 1 | 1 | 1 | 2

9. Secondary Outcome: Number of Participants With Solicited Systemic Reactions Occurring Within 7 Days of Booster Vaccination
Description: Participants were monitored for systemic reactions from 30 minutes through 7 days post booster vaccination. Systemic reactions (general signs / symptoms) included the following:
  * Fever
  * Change in eating habits
  * Diarrhea
  * Sleepiness
  * Irritability
  * Unusual crying
  * Vomiting
  Fever was graded as follows:
  * Grade 1: 37.5 ℃ to 37.9 ℃
  * Grade 2: 38.0 ℃ to 38.4 ℃
  * Grade 3: 38.5 ℃ to 40.0 ℃
  * Grade 4: > 40.0 ℃
  Change in eating habits, diarrhea, sleepiness, irritability, unusual crying, vomiting were graded as follows:
  * Grade 1: causing no or minimal interference with usual social or functional activities
  * Grade 2: causing greater than minimal interference with usual social or functional activities
  * Grade 3: causing inability to perform usual social or functional activities OR hospitalization indicated
  * Grade 4: inability to perform basic self-care OR medical or operative intervention indicated to prevent permanent impairment, persistent disability, or death.
Time Frame: From 30 minutes to 7 days following booster vaccination (Study Day 365 to 372)
Population: Participants who received the booster vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | Group A: CD-JEV | Group B: CD-JEV | Total
Number analyzed (Participants) | 424 | 109 | 533
Participants
  Any systemic reaction | 14 | 5 | 19
  Fever | 10 | 3 | 13
  Fever - Grade 1 | 8 | 3 | 11
  Fever - Grade 2 | 4 | 0 | 4
  Change in eating habits | 1 | 1 | 2
  Change in eating habits - Grade 1 | 1 | 1 | 2
  Diarrhea | 0 | 0 | 0
  Sleepiness | 0 | 0 | 0
  Irritability | 1 | 0 | 1
  Irritability - Grade 1 | 1 | 0 | 1
  Unusual crying | 0 | 0 | 0
  Vomiting | 2 | 1 | 3
  Vomiting - Grade 1 | 2 | 1 | 3

10. Secondary Outcome: Number of Participants With Unsolicited Adverse Events (AEs) and Serious Adverse Events (SAEs) Within 28 Days Following Booster Vaccination
Description: AEs were graded for severity according to the following:
  Grade 1 (Mild): Symptoms causing no or minimal interference with usual social and functional activities
  Grade 2 (Moderate): Symptoms causing greater than minimal interference with usual social and functional activities
  Grade 3 (Severe): Symptoms causing inability to perform usual social and functional activities with intervention or hospitalization indicated
  Grade 4 (Potentially life-threatening): Symptoms causing inability to perform basic self-care functions OR medical or operative intervention indicated to prevent permanent impairment, persistent disability, or death.
  Relationship to study vaccine was based on the Clinician's assessment.
  A serious adverse event is defined as an AE that meets 1 of the following criteria:
  * Death
  * Life-threatening
  * Requires hospitalization or prolongation of existing hospitalization
  * Results in persistent disability
  * Important medical event based on medical judgement
Time Frame: 28 days following booster vaccination (Study Days 365 to 393)
Population: Participants who received the booster vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | Group A: CD-JEV | Group B: CD-JEV | Total
Number analyzed (Participants) | 424 | 109 | 533
Participants
  Any adverse events | 57 | 26 | 83
  Mild adverse events | 48 | 22 | 70
  Moderate adverse events | 8 | 4 | 12
  Severe adverse events | 1 | 0 | 1
  Life-threatening adverse events | 0 | 0 | 0
  Related adverse events | 3 | 1 | 4
  Unrelated adverse events | 54 | 25 | 79
  Serious adverse events | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 28 days after booster vaccination (Study Day 365 to 393)
Description: Adverse events are reported for all participants who received the CD-JEV booster vaccination.
Arm/Group | Group A: CD-JEV | Group B: CD-JEV | Total
All-Cause Mortality (participants affected / at risk) | 0/424 | 0/109 | 0/533
Serious Adverse Events (participants affected / at risk) | 0/424 | 0/109 | 0/533
Other Adverse Events (participants affected / at risk) | 57/424 | 26/109 | 83/533
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group A: CD-JEV (N=424) | Group B: CD-JEV (N=109) | Total (N=533)
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 1
Otorrhoea (Ear and labyrinth disorders) | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 1
Toothache (Gastrointestinal disorders) | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 4 | 1 | 5
Injection site pain (General disorders) | 1 | 0 | 1
Pain (General disorders) | 0 | 1 | 1
Pyrexia (General disorders) | 10 | 1 | 11
Acarodermatitis (Infections and infestations) | 2 | 2 | 4
Cellulitis (Infections and infestations) | 1 | 0 | 1
Conjunctivitis (Infections and infestations) | 0 | 3 | 3
Dysentery (Infections and infestations) | 3 | 1 | 4
Furuncle (Infections and infestations) | 2 | 0 | 2
Gastroenteritis (Infections and infestations) | 1 | 0 | 1
Measles (Infections and infestations) | 1 | 0 | 1
Mumps (Infections and infestations) | 3 | 0 | 3
Nasopharyngitis (Infections and infestations) | 2 | 4 | 6
Otitis media (Infections and infestations) | 1 | 0 | 1
Pharyngitis (Infections and infestations) | 1 | 1 | 2
Respiratory tract infection (Infections and infestations) | 1 | 0 | 1
Rhinitis (Infections and infestations) | 2 | 0 | 2
Skin infection (Infections and infestations) | 0 | 1 | 1
Subcutaneous abscess (Infections and infestations) | 0 | 1 | 1
Tonsillitis (Infections and infestations) | 1 | 1 | 2
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 1
Urinary tract infection (Infections and infestations) | 3 | 0 | 3
Animal scratch (Injury, poisoning and procedural complications) | 0 | 1 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 2 | 2
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Gastric pH decreased (Investigations) | 1 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 1
Headache (Nervous system disorders) | 1 | 0 | 1
Irritability (Psychiatric disorders) | 1 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 2 | 7
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 7 | 3 | 10
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Lower respiratory tract infection (Gastrointestinal disorders) | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-03-04): https://cdn.clinicaltrials.gov/large-docs/46/NCT02514746/Prot_000.pdf
  • Statistical Analysis Plan (2018-07-12): https://cdn.clinicaltrials.gov/large-docs/46/NCT02514746/SAP_001.pdf